CLINICAL TRIAL: NCT05462132
Title: A Phase 1, Dose-escalation, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacodynamics of SYNB1353 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacodynamics of SYNB1353 in Healthy Adult Volunteers
Acronym: HCU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SYNB1353-CP-001
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Homocystinuria
Keywords: HCU; Amino acid metabolism; Inborn error of metabolism
MeSH Terms: conditions — Homocystinuria; Metabolism, Inborn Errors

STUDY DESIGN:
Intervention Model Description: Dose-escalation decisions will be made once at least 6 subjects in a cohort have received IMP and have had at least 24 hours of post-dose observation. Dose escalation will be up to approximately 3-fold per cohort.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Decisions will be made based on a blinded review of tolerability, clinical observations, safety laboratory assessments, and, optionally, PD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): HV subjects receive doses 3 × 10^11 live cells of SYNB1353 and 30 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of 30 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 2 (Experimental): HV subjects receive doses 3 × 10^11 live cells of SYNB1353 and up to 100 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of up to 100 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 3 (Experimental): HV subjects receive doses 6 × 10^11 live cells of SYNB1353 and 30 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of 30 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 4 (Experimental): HV subjects receive doses 6 × 10^11 live cells of SYNB1353 and up to 100 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of up to 100 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 5 (Experimental): HV subjects receive doses 1 × 10^12 live cells of SYNB1353 and 30 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of 30 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 6 (Experimental): HV subjects receive doses 1 × 10^12 live cells of SYNB1353 and up to 100 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of up to 100 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 7 (Experimental): HV subjects receive doses less than or equal to 2 × 10^12 live cells of SYNB1353 and 30 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of 30 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353
- Cohort 8 (Experimental): HV subjects receive doses less than or equal to 2 × 10^12 live cells of SYNB1353 and up to 100 mg/kg of methionine.
  Subjects will receive a single dose of SYNB1353 on the first day of dosing (Day 1), on Days 2 and 3 subjects will receive up to 2 doses of IMP (BID), and on Days 4 to 7 subjects will receive up to 3 doses of IMP (TID).
  A methionine loading study will be performed on Day -1 and Day 7 after an overnight fast. A dose of methionine of up to 100 mg/kg will be evaluated.
  Interventions: Drug: SYNB1353

INTERVENTIONS:
Drug: SYNB1353 — SYNB1353 IMP is formulated as a nonsterile solution intended for oral administration. SYNB1353 is subsequently lyophilized to form the bulk drug product. The lyophilized product is sieved into powder form and filled into high-density polyethylene (HDPE) bottles. Placebo will be manufactured using an inactive powder that is color matched to the SYNB1353 drug product. L-Methionine will be supplied as dry powder and will be suspended in a diluent prior to use.

SUMMARY:
This is a Phase 1, double-blind (Sponsor-open), placebo-controlled, randomized, dose-escalation, inpatient study using a multiple-ascending dose (MAD) design to assess the safety, tolerability, and PD of SYNB1353 in HVs.

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability and PD of SYNB1353 in up to 8 cohorts of HVs. In each cohort, HVs will be randomly assigned to investigational medicinal product (IMP), according to a MAD design, to receive either SYNB1353 or placebo (6 active:2 placebo per cohort). A methionine loading study will be performed on Day -1 and Day 7. At each IMP dose level, a dose of methionine will be evaluated. The methionine dose may increase if necessary to evaluate the PD of SYNB1353.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to ≤ 64 years.
2. Able and willing to voluntarily complete the informed consent process.
3. Available for and agree to all study procedures, including feces, urine, and blood collection and adherence to diet control, inpatient monitoring, follow-up visits, and compliance with all study procedures.
4. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as a condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion # 5) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the IMP.
5. Female subjects who meet 1 of the following:

   1. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (human chorionic gonadotropin) at Screening and a negative urine pregnancy test at baseline prior to the start of IMP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion # 4) after informed consent, throughout the study and for a minimum of 3 months after the last dose of IMP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, and/or vasectomized partner with documented azoospermia 3 months after procedure.
   2. WOCBP must not be breastfeeding.
   3. Premenopausal women with at least 1 of the following:

   i. Documented hysterectomy ii. Documented bilateral salpingectomy iii. Documented bilateral oophorectomy iv. Documented tubal ligation/occlusion v. Sexual abstinence is preferred or usual lifestyle of the subject d. Postmenopausal women (12 months or more amenorrhea verified by follicle- stimulating hormone [FSH] assessment and over 45 years of age in the absence of other biological or physiological causes).

Exclusion Criteria:

1. Acute or chronic medical, surgical, psychiatric, or social condition or laboratory abnormality that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of study safety or PD results and, in the judgment of the Investigator, would make the subject inappropriate for enrollment.
2. Body mass index < 18.5 or ≥ 35 kg/m2.
3. History of or current immunodeficiency disorder including human immunodeficiency virus (HIV) antibody positivity.
4. Hepatitis B surface antigen positivity (subjects with hepatitis B surface antibody positivity and hepatitis B core antibody positivity are not excluded, provided that the hepatitis B surface antigen is negative).
5. Hepatitis C antibody positivity, unless a hepatitis C virus ribonucleic acid test is performed, and the result is negative.
6. History of febrile illness, confirmed bacteremia, or other active infection deemed clinically significant by the Investigator within 30 days prior to the anticipated first dose of IMP.
7. History of (within the past month) passage of 3 or more loose stools per day, where "loose stool" is defined as a Type 6 or Type 7 on the Bristol Stool Chart (see Appendix 1).
8. Inflammatory or irritable bowel disorder of any grade experienced within the previous 60 days.
9. Active or past history of GI bleeding within 60 days prior to the Screening Visit as confirmed by hospitalization-related event(s) or medical history of hematemesis or hematochezia.
10. Underlying cardiovascular disease or uncontrolled gastroesophageal reflux disease
11. Intolerance of or allergic reaction to EcN, esomeprazole and all other PPIs, or any of the ingredients in SYNB1353 or placebo formulations.
12. Allergy or intolerance to multiple antibiotics which would preclude use of antibiotics for eradication of SYNB1353 in case of colonization.
13. Currently taking or plans to take Methotrexate, Azuridine, Nitrous Oxide, Phenytoin, or Carbamazepine.
14. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 28 days prior to the first anticipated dose of IMP through final assessment, including planned surgery, hospitalizations, dental procedures, or interventional studies that are expected to require antibiotics. Exception: topical antibiotics are allowed.
15. Major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay within the past 3 months prior to Screening.
16. Dependence on alcohol or drugs of abuse.
17. Administration or ingestion of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the Screening Visit, or current enrollment in an investigational study.
18. Screening laboratory parameters (e.g., chemistry panel, hematology, coagulation) and ECG outside of the normal limits based on standard ranges or as judged to be clinically significant by the Investigator. A single repeat evaluation is acceptable.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal laboratory values and/or adverse events | Day -2 through Day 8
  Lab results outside of the central laboratory normal range parameters will be considered abnormal and reviewed for clinical significance and reported as AEs. AEs will be evaluated using the NCI CTCAE v5.0

SECONDARY OUTCOMES:
The rate at which the SYNB1353 strain clears | Up to 14 weeks following the last dose of IMP
  Clearance is measured in feces by quantitative polymerase chain reaction (qPCR). A negative in fecal SYNB1353 qPCR is defined as a result below the limit of quantification.

CONTACTS AND LOCATIONS:
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No